CLINICAL TRIAL: NCT04236960
Title: Phase I Clinical Study of Meningococcal Group ACYW135 Conjugate Vaccine
Brief Title: Safety Evaluation of Meningococcal Group ACYW135 Conjugate Vaccine in 2-month to 55 Years Old Population.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Walvax Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 008152017002
Record Dates: First submitted 2018-07-05; First posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Meningococcal Infections
Keywords: Meningitis, Meningococcal, Serogroup A; Meningitis, Meningococcal, Serogroup C; Meningitis, Meningococcal, Serogroup Y; Meningitis, Meningococcal, Serogroup W135
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 18~55 yrs (Experimental): 1 dose of meningococcal group ACYW135 conjugate vaccine will be administered on day 0.
  Interventions: Biological: Meningococcal Group ACYW135 Conjugate Vaccine
- 2~17 yrs (Experimental): 1 dose of meningococcal group ACYW135 conjugate vaccine will be administered on day 0.
  Interventions: Biological: Meningococcal Group ACYW135 Conjugate Vaccine
- 7~23 mos (Experimental): 2 doses of meningococcal group ACYW135 conjugate vaccine will be administered. One-month interval between the first and second dose.
  Interventions: Biological: Meningococcal Group ACYW135 Conjugate Vaccine
- 3 mos (Experimental): 3 doses of meningococcal group ACYW135 conjugate vaccine will be administered. One-month interval between every two doses.
  Interventions: Biological: Meningococcal Group ACYW135 Conjugate Vaccine
- 2 mos (Experimental): 3 doses of meningococcal group ACYW135 conjugate vaccine will be administered. Two-month interval between every two doses.
  Interventions: Biological: Meningococcal Group ACYW135 Conjugate Vaccine

INTERVENTIONS:
Biological: Meningococcal Group ACYW135 Conjugate Vaccine — 1 dose in Stage 1 (2~55 yrs), 2 doses in Stage 2 (7~23 mos), and 3 doses in Stage 3 (2&3 mos)

SUMMARY:
A single-center and open-labeled Phase I study, designed to evaluate the safety by observing the occurrence of adverse events and change of hematology, liver and renal function after vaccination of a meningococcal group A, C, Y, and W135 conjugate vaccine in healthy population aged 2 months to 55 years old.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children, adolescents and adults (age range: 2 months to 55 years old) based on medical history, physical examination or judgement of the investigator
* Subjects aged ≥18 years old voluntarily agree to participate in this clinical study and sign the informed consent form; or for subjects aged <18 years old, the legal guardian voluntarily agrees that his/her child to participate in this clinical study, and sign the informed consent form. For juveniles aged ≥8 years old, both the subject and his/her legal guardians should voluntarily agree to participate in this clinical study and sign the informed consent form.
* The subject and his/her legal guardians as well as the family members are able to follow the request of clinical study protocol.
* Subjects aged 2 or 3 months should have no vaccination history of any meningococcal vaccine; subjects aged 7~23 months should have not received any other meningococcal vaccine except the meningococcal group A polysaccharide vaccine included in National Immunization Program, and the time since last vaccination of meningococcal group A polysaccharide vaccine should be >6 months; for subjects ≥2 years, the time since last vaccination of meningococcal vaccine should be >2 years.
* For subjects aged ≥2 years, there should be no clinically significant abnormal hematology, liver and renal function results judged by the investigator before immunization.
* Subjects should not receive any attenuated live vaccine 14 days, or inactivated vaccine 7 days before or after vaccination.
* Axillary temperature ≤37.0℃.

Exclusion Criteria for First Dose:

* Subjects aged 2 or 3 months at enrollment with birth weight <2.5 kg.
* Subjects aged 2 or 3 months at enrollment had received blood products and immunoglobin after birth; subjects of other age groups had received blood products or immunoglobin in <3 months before vaccination.
* Subjects aged <12 months at enrollment are diagnosed as with pathological jaundice or have a history of pathological jaundice.
* Subjects aged <2 months at enrollment had abnormal labor (dystocia, assisted instrumental delivery) or with the history of asphyxia or nervous damage.
* Subjects aged ≥18 years who are planning pregnancy, or are pregnant, or are breastfeeding.
* Subjects aged ≥18 years with uncontrollable hypertension (during screening: systolic BP >140 mmHg or diastolic BP >90 mmHg).
* Subjects are known to be allergic to certain components contained in the investigational vaccine (mainly include: capsular polysaccharide of meningococcal group A, group C, group Y, or group W135, diphtheria toxoid or diphtheria antigen).
* Subjects with the history of serious allergy to any vaccine or drug. (including but not limited to: allergic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, local allergic necrosis reaction [Arthus reaction]).
* Subjects with the history of meningitis.
* Subjects with moderate to severe fever (axillary temperature ≥38.0℃) in last 3 days.
* Subjects with the history or family history of convulsion, seizure, encephalopathy, or psychiatric disorders.
* Subjects with definite diagnosis of thrombocytopenia or other coagulation disorders.
* Subjects with primary or secondary immunological dysfunction, including HIV infection, disorder or resection of thyroid, pancreas, liver, spleen or kidney; or needed treatment due to thyroid disorders in last 12 months (time interval <12 months).
* Subjects have received immunosuppressive therapy, cytotoxic therapy, corticosteroid hormone (not include corticosteroid hormone spray for allergic rhinitis, epithelial corticosteroid hormone for acute and non-complicated dermatitis) in last 6 months (time interval <6 months).
* Subjects with known congenital malformation, developmental disabilities or clinically confirmed serious chronic diseases (e.g., Down syndrome, diabetes mellitus, sickle cell anemia or nervous disease, Guillain-Barre syndrome, etc.).
* Subjects with known or suspected diseases that are likely to affect the vaccination by investigators' judgement, such as: serious respiratory diseases, acute infection or the active period of chronic disease, serious cardiovascular diseases, liver and renal diseases, malignant tumors, serious infectious or allergic skin diseases.
* Subjects are participating or plan to participate in other clinical trials of investigational medications.
* Any other conditions that may influence the evaluation of clinical study by investigators' judgement.

Exclusion Criteria for Second and Third Dose:

* New conditions that conforms with the exclusion criteria for first dose.
* Subjects that develop grade 4 adverse reactions after vaccination of investigational vaccine.
* Subjects that develop serious allergic reactions after vaccination of investigational vaccine.
* Any other conditions that may influence the evaluation of clinical study by investigators' judgement based on the exclusion criteria for first dose.

Ages: 2 Months to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2019-11-28 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events after each vaccination | 30 days after vaccination
  Percentage of subjects with local and systemic adverse events after each dose of vaccination

SECONDARY OUTCOMES:
Incidence of serious adverse events after vaccination | day 0 to 6 months after last dose
  Percentage of subjects with serious adverse events from day 0 to 6 months after last dose
Blood routine in 2 years and above subjects | 3 days after vaccination
  content of hemoglobin（g/dL）、white blood cell count（WBC）、blood platelet count（PLT）3 days after vaccination in 2 years and above subjects
Liver function in 2 years and above subjects | 3 days after vaccination
  Alanine aminotransferase（ALT），Aspartate aminotransferase（AST），Total bilirubin(TBIL) 3 days after vaccination in 2 years and above subjects
Renal function in 2 years and above subjects | 3 days after vaccination
  Creatinine（CR），Urea nitrogen（BUN）3 days after vaccination in 2 years and above subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial Center for Disease Control and Prevention, Guangzhou, Guangdong, China